CLINICAL TRIAL: NCT00407082
Title: A Multicenter, Randomized, Double-Masked, Controlled Study to Evaluate the Safety & Efficacy of Intravitreal Fluocinolone Acetonide (0.59 or 2.1 mg) Implant in Subjects With Non-Infectious Uveitis Affecting the Posterior Segment of the Eye
Brief Title: Safety and Efficacy of Fluocinolone Acetonide Intravitreal Implants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 415-001
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Noninfectious Posterior Uveitis
MeSH Terms: interventions — Fluocinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluocinolone acetonide 0.59mg (Experimental): Fluocinolone acetonide ocular implant 0.59mg
  Interventions: Drug: fluocinolone acetonide intravitreal implant
- Fluocinolone acetonide 2.1mg (Experimental): Fluocinolone acetonide ocular implant 2.1mg
  Interventions: Drug: Fluocinolone acetonide 2.1mg
- No intervention (No Intervention): Fellow eye

INTERVENTIONS:
Drug: fluocinolone acetonide intravitreal implant — Fluocinolone acetonide ocular implant 0.59mg
  Arms: Fluocinolone acetonide 0.59mg
Drug: Fluocinolone acetonide 2.1mg — Fluocinolone acetonide ocular implant 2.1mg
  Arms: Fluocinolone acetonide 2.1mg

SUMMARY:
This is a multi-center, randomized, double-masked, controlled study to evaluate the safety and efficacy of fluocinolone acetonide (FA) intravitreal implants for the management of subjects with non-infectious uveitis affecting the posterior segment of the eye. An additional objective is to compare the safety and efficacy of two doses of fluocinolone acetonide.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females at least 6 years of age who had been diagnosed and treated for recurrent, non-infectious uveitis affecting the posterior segment of one or both eyes for at least 1 year prior to the start of the study, and had 'quiet' eyes at surgery

Exclusion Criteria:

* Coexisting medical or ocular conditions that would interfere with the study results

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2000-12; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Recurrence of uveitis before and after implantation. | 34 weeks pre-implantation; 34 weeks, 1 year, 2 years and 3 years post-implantation

SECONDARY OUTCOMES:
Post-implantation rate of uveitis recurrence, within patient comparison of implanted vs fellow eyes. | 34 weeks, 1 year, 2 years and 3 years post-implantation
Post-implantation time to recurrence of uveitis within patient comparison of implanted vs fellow eyes. | 34 weeks, 1 year, 2 years and 3 years post-implantation
The need for adjunctive uveitis treatment for the study eye, within patient comparison (pre- versus post-implantation) | 34 weeks, 1 year, 2 years and 3 years post-implantation
Reduction in the area of cystoid macular edema (CME) within patient comparison of responding eyes (implant vs fellow eyes) | 34 weeks, 1 year, 2 years and 3 years post-implantation
Results of QOL surveys pre- versus post-implantation | 34 weeks, 1 year, 2 years and 3 years post-implantation
Visual acuity, within patient comparison of responding eyes (implant vs fellow eyes) | 34 weeks, 1 year, 2 years and 3 years post-implantation
Time to recurrence, between treatment group comparison | 34 weeks, 1 year, 2 years and 3 years post-implantation
Post implantation uveitis rate, between treatment group comparison | 34 weeks, 1 year, 2 years and 3 years post-implantation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Crescuillo, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Jaffe GJ, Martin D, Callanan D, Pearson PA, Levy B, Comstock T; Fluocinolone Acetonide Uveitis Study Group. Fluocinolone acetonide implant (Retisert) for noninfectious posterior uveitis: thirty-four-week results of a multicenter randomized clinical study. Ophthalmology. 2006 Jun;113(6):1020-7. doi: 10.1016/j.ophtha.2006.02.021. Epub 2006 May 9. PMID 16690128
- [Derived] Callanan DG, Jaffe GJ, Martin DF, Pearson PA, Comstock TL. Treatment of posterior uveitis with a fluocinolone acetonide implant: three-year clinical trial results. Arch Ophthalmol. 2008 Sep;126(9):1191-201. doi: 10.1001/archopht.126.9.1191. PMID 18779477